CLINICAL TRIAL: NCT01134302
Title: The Influence of Postoperative Systemic Oxygen Transport on Neurologic and Functional Outcomes in Infants Undergoing Single Ventricle Palliation With Norwood and Hybrid Management Strategies
Brief Title: Hybrid Versus Norwood Management Strategies in Infants Undergoing Single Ventricle Palliation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Christopher Caldarone, Principal Investigator, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1000013962
Record Dates: First submitted 2010-03-23; First posted 2010-05-31 (Estimated); Last update posted 2010-05-31 (Estimated); Status verified 2010-05

CONDITIONS: Congenital Heart Disease
Keywords: Hybrid; Norwood; congenital heart disease; single ventricle
MeSH Terms: conditions — Heart Defects, Congenital; Univentricular Heart

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Active Comparator): Hybrid Management
  Interventions: Procedure: Hybrid Strategy
- Arm 2 (Active Comparator): Norwood Management
  Interventions: Procedure: Norwood management strategy

INTERVENTIONS:
Procedure: Norwood management strategy — Norwood palliation will be performed as per current clinical practice at The Hospital for Sick Children.
  Arms: Arm 2
Procedure: Hybrid Strategy — Hybrid palliation will be performed as per current clinical practice at The Hospital for Sick Children.
  The 'Hybrid' management strategy utilizes catheter-based and non-open heart surgical procedures in the neonatal period to stabilize the neonate.10 The majority of the reconstruction is thereby deferred to 4-6 months of age, at which time the second stage procedure including an aortic arch reconstruction is performed. The third stage procedure (Fontan) is identical between Norwood and Hybrid strategies.
  Arms: Arm 1

SUMMARY:
The purpose of this trial is to determine, at 3 years of life, how the neurologic and functional outcomes in infants with single ventricles are different when comparing children treated with the Hybrid strategy to the Norwood strategy.

DETAILED DESCRIPTION:
Neurologic deficits in children with single ventricle physiology are believed to be associated with the reconstruction of the aortic arch during the initial Norwood procedure as a neonate. In the last few years, a new management strategy (the 'Hybrid' strategy) has been proposed which defers the aortic arch reconstruction to a second stage procedure at 4-6 months of age.

Proponents of the Hybrid strategy assert that the avoidance of cardiopulmonary bypass and circulatory arrest in the neonatal period will avoid neurologic injury in the critical neonatal period and thereby result in superior long-term neurologic outcomes.

We are testing whether the Hybrid management strategy is associated with superior neurologic outcomes or not.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of functional single ventricle anatomy amenable to Norwood or Hybrid first stage palliation.
2. Informed consent of parent(s) or legal guardian.

Exclusion Criteria:

1. Pre-operative identification of anatomy rendering either a Norwood or Hybrid procedure clinically inappropriate;
2. Recent history of significant cerebral bleed or necrotizing enterocolitis;
3. Severe hemodynamic instability;
4. Any other major congenital abnormality (i.e. congenital diaphragmatic hernia, tracheoesophageal fistula) or clinically significant acquired extra-cardiac disorder (e.g. meconium aspiration with need for high frequency ventilation, persistent renal failure requiring dialysis).

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Neurologic and functional outcomes | 14 months of age
  Neurodevelopmental and functional status will be assessed at 14 months of age using the Bayley Scales of Infant Development®-Third Edition (BSID-III), MacArthur Commmunicative Development Inventory/Words and Gestures (CDI) and Functional Status-II-Revised Questionnaire.
Neurologic and functional outcomes | 3 years of age (during procedure 3 pre-op)
  At ~3 years of age, the Vineland Scale,the Mullen Developmental Scale, and the BASC behavioural scale will be formally assessed

SECONDARY OUTCOMES:
Hemodynamic Assessment | Baseline and 4-6 months
  Arterial, superior vena cava and pulmonary vein pressure will be monitored via indwelling catheters. This measurement will be taken during: procedure 1 pre-op, procedure 1 post-op, procedure 2 pre-op, and procedure 2 post-op.
Blood Sampling | Baseline and 4-6 months
  Standard blood gas samples will be drawn from indwelling arterial, SVC and pulmonary vein catheters to provide oxygen saturation and lactate data. This measurement will be taken immediately after chest opening, and then postoperatively at 2 hour intervals during the first 24 hours and at 4 hour intervals during the following 48 hours after first and second stage procedures.
Systemic Oxygen Consumption | Baseline and 4-6 months
  Measurement of pre- and post-operative VO2. This measurement will be taken during: procedure 1 pre-op, procedure 1 post-op, and procedure 2 pre-op
Cerebral Oxygen Transport Surrogate Measurements | Baseline and 4-6 months
  Cerebral oxygen saturation (ScO2) will be continuously measured by Near Infrared Spectroscopy (NIRS). This measurement will be taken during: procedure 1 pre-op, procedure 1 post-op, procedure 2 pre-op, and procedure 2 post-op.
Cerebral Blood Flow Velocity | Baseline and 4-6 months
  Transcranial Doppler sonography using the TCD through the middle cerebral artery with a 2 MHz pulse-wave ultrasound transducer will be used to measure cerebral blood flow velocity non-invasively.
  This measurement will be taken during: procedure 1 pre-op, procedure 1 post-op, procedure 2 pre-op, and procedure 2 post-op.
Electroencephalograph | Baseline and 4-6 months
  Locked digital video electroencephalography (DVEEG) will be used to continuously monitor ischemic injury and seizures. This will be done at the folling times: procedure 1 pre-op, procedure 1 post-op prior to discharge, and procedure 2 post-op.
MRI scans | Baseline, 4-6 months and 2-3 years
  Brain imaging will be assessed for evidence of congenital malformations or structural abnormalities, cerebral edema, acute ischemia, intracranial hemorrhages, periventricular leukomalacia (PVL), focal tissue loss, atrophy, delays in myelin maturation and infarcts.
  The MRI will be done during procedure 1 post-op prior to discharge, procedure 2 post-op prior to discharge and procedure 3 pre-op.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Caldarone, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- See also: Related Info — http://www.sickkids.ca/Centres/heart-centre/index.html
- See also: Related Info — http://www.ctsnet.org/home/gvanarsdell
- See also: Related Info — http://www.sickkids.ca/Research/REB/index.html